CLINICAL TRIAL: NCT05201586
Title: Conditional Cash Transfers to Address Social Determinants of Health and Social Needs in a Primary Care Clinic
Brief Title: CCTs to Address Social Needs in a Primary Care Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 849553
Record Dates: First submitted 2021-10-15; First posted 2022-01-21 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Health-Related Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conditional cash transfer (Active Comparator): Investigators will randomize 15 patients into this intervention arm. All participants will undergo a semi-structured patient interview about how social needs impact health and self-perceptions of health at the time of enrollment and again in 6 months. All participants will receive a CCT after the first interview.
  Interventions: Other: Conditional Cash Transfer; Other: Semi-structured interviews
- Control (Active Comparator): Investigators will randomize 15 patients into this control arm. All participants will undergo a semi-structured patient interview about how social needs impact health and self-perceptions of health at the time of enrollment and again in 6 months.
  Interventions: Other: Semi-structured interviews

INTERVENTIONS:
Other: Conditional Cash Transfer — CCTs will be given to participants in the form of a pre-loaded debit card.
  Arms: Conditional cash transfer
Other: Semi-structured interviews — Research team will conduct semi-structured interviews exploring how social determinants of health and social needs impact health. Participants will be asked to set a health goal. 6 months after the initial interview, the team will interview the patients again and evaluate whether that health goal was achieved.

SUMMARY:
This is a study of conditional cash transfers (CCTs) to address social needs impacting the health of low-income patients in West Philadelphia who screen positive for financial strain, transportation needs, or food insecurity. Participants will be randomized to receive a CCT at enrollment. All participants will be interviewed at time of enrollment and again in 6 months to investigate if a CCT affected objective health outcomes, individual health goals, and self-rated perceptions of health.

DETAILED DESCRIPTION:
This is a randomized trial of the effect of conditional cash transfers (CCTs) on West Philadelphia residents who are patients at two Division of General Internal Medicine primary care clinics located at 3701 Market Street. Currently, our practice administers social determinants of health (SDOH) screening questionnaires which are available to review as part of a patients electronic medical record. Eligible patients will have been flagged as having at least 1 of 3 social needs: financial resource strain, transportation needs, and food insecurity. From this pool, patients with Medicare and Medicaid insurance who live in low income neighborhoods in Philadelphia will be recruited. Eligible participants will be older than 18 years old with at least 1 chronic medical condition including obesity, diabetes, hypertension, chronic kidney disease, coronary artery disease, chronic lung disease, active smoker, and stroke. Eligible patients will be randomized to either the CCT arm or control. Verbal consent will be obtained from all participants allowing the study team to collect personal health information and conduct audio-recorded semi-structured patient interviews. Personal health information will include demographics, chronic medical conditions, weight, blood pressure, cigarettes per day, and last hemoglobin A1c. Utilization outcomes such as ED visits, hospital admissions, and primary care office visits using Epic will be recorded. This data will be collected in REDCap at the time of enrollment and at the end of the 6-month study period. Patient interviews will be conducted by a research assistant. The participants will have the option of conducting the interviews in-person using a private room within the primary care clinic or virtually using a secure telehealth platform. Translation services will be provided, if needed. The patient will first complete the Short Form-12 (SF-12) survey, a validated multidimensional generic measure of health-related quality of life. For interviews conducted in-person, a paper version of the SF-12 will be given to the patients and collected at the end of the interview. For interviews conducted virtually, the interviewer will orally present the SF-12 survey to the participant and record the answers in a paper format. The interviewer will then conduct an audio-recorded semi-structured enrollment interview exploring patient perceptions about the social need flagged in the SDOH screening questionnaire, how it impacts health, and asked to set a personal health goal to achieve over the next 6 months. Participants who were randomized to receive the CCT will be asked to use it towards the SDOH risk factor flagged by the social needs assessment. If the patient chooses to spend money on something not related to identified social need, there will be no punitive financial repercussions or payback required. The CCT will be given in the form of a pre-loaded electronic debit card like the Clincard. The study team will not review expenses of participants during or after the study is complete. Six months after the initial interview, all participants will again complete the SF-12 survey and the research assistant will conduct audio-recorded semi-structured exit interviews either in-person or virtually. These interviews will explore whether the patients achieved their health goal. Participants who received the CCT will be asked additional questions exploring whether the CCT helped achieve that goal. At the end of each interview, audio tapes will be sent for external transcription by a HIPAA compliant transcription service and then analyzed with the help of the research assistant working with the study team.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be 18-89 years old of any gender
* At least 1 chronic medical condition including obesity, diabetes, hypertension, chronic kidney disease, coronary artery disease, chronic lung disease, active smoker, and stroke.
* Participants with Medicare and/or Medicaid insurance
* Home address falls within a West Philadelphia zip code (19104, 19131, 19139, 19143, 19151)

Exclusion Criteria:

* Adults 90 and older
* Patients who are unable to provide consent due to mental disability or illness
* Patients unable to participate in a verbal interview due to a physical or mental health condition will also be excluded

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Themes in interview data | 6 months
  The primary outcome is to identify main themes in the interview data of how social needs impact health and what effect CCTs may have have on patient perceptions of health. The audio recordings will be sent for external transcription by a HIPAA compliant transcription service. The transcriptions will be coded and analyzed in nVivo, a qualitative data management system. Content analyses will be used to discover the main themes in the interview data and then look at associations among the prevalence of themes and social needs within and between groups.

SECONDARY OUTCOMES:
Short Form (SF)-12 survey | 6 months
  Interviews will include administration of an SF-12 survey and a secondary outcome will look at differences in SF-12 answers between groups before and after intervention. The SF-12 is a validated health-related quality-of-life questionnaire consisting of twelve questions that assess patient's perceptions of physical and mental health. The SF-12 does not use a scoring scale; answers consist instead of "yes, no" or ratings of "not at all, a little bit, moderately, quite a bit, or extremely."
Objective health metrics - Blood pressure | 6 months
  Most recent available blood pressure will be documented at the time of enrollment and again in 6 months. Changes to these clinical measures will be investigated between the control and intervention groups.
Objective health metrics - Hemoglobin A1c | 6 months
  Most recent available diabetes number or Hemoglobin A1c will be documented at the time of enrollment and again in 6 months. Changes to these clinical measures will be investigated between the control and intervention groups.
Objective health metrics - Cigarettes per day | 6 months
  If patient smokes, the number of cigarettes per day will be documented at the time of enrollment and again in 6 months. Changes to these clinical measures will be investigated between the control and intervention groups.
Utilization data - Emergency department (ED) visits | 6 months
  The number of emergency department (ED) visits of each participant in the 6 months before enrollment and during the study period will be documented. Changes to these clinical measures will be investigated between the control and intervention groups.
Utilization data - Hospital admissions | 6 months
  The number of hospital admissions of each participant in the 6 months before enrollment and during the study period will be documented. Changes to these clinical measures will be investigated between the control and intervention groups.
Utilization data - Primary Care Office Visits | 6 months
  The number of primary care office visits of each participant in the 6 months before enrollment and during the study period will be documented. Changes to these clinical measures will be investigated between the control and intervention groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No